CLINICAL TRIAL: NCT00600158
Title: Effects of Intravenous Local Anesthetic on Bowel Function After Colectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Marcel E. Durieux, MD PhD, Professor of Anesthesiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED001
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Postoperative Ileus
Keywords: colectomy
MeSH Terms: interventions — Bupivacaine; Hydromorphone; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): lidocaine intravenously
  Interventions: Drug: lidocaine
- 1 (Active Comparator): epidural local anesthetic
  Interventions: Drug: bupivacaine with hydromorphone

INTERVENTIONS:
Drug: bupivacaine with hydromorphone — bupivacaine 0.125% with hydromorphone 6 mcg/ml epidurally at 10 ml/h
  Arms: 1
Drug: lidocaine — lidocaine 2 mg/min intravenously (or 3 mg/kg in patients > 70 kg)
  Arms: 2

SUMMARY:
Epidural local anesthetics are the gold standard for shortening duration of bowel dysfunction after bowel surgery. Previous studies suggest that their effect may be in part a result of actions of the local anesthetic outside the epidural space. If local anesthetics could be administered intravenously instead, this might be a safer, easier and less expensive approach. Therefore, this trial will compare the effect on bowel function recovery of intravenous local anesthetics with those administered epidurally.

DETAILED DESCRIPTION:
Ileus seems an almost unavoidable side effect of most types of bowel surgery. This is unfortunate, since postoperative ileus is not only unpleasant for the patient, but also has detrimental effects on recovery from surgery. The maintenance of enteral nutrition has been shown to be an important factor in ensuring rapid recovery from gastrointestinal surgery, as the catabolic state decreases immune function, delays wound healing, and increases morbidity. However, ileus often precludes enteral feeding. As a result, duration of postoperative ileus is frequently a major determinant of duration of hospitalization. At this time, the most effective manner to minimize the duration of postoperative ileus is the use of continuous local anesthetic epidural analgesia 3 as confirmed by a systematic review on the topic. This effect appears specifically related to the use of local anesthetic, as postoperative epidural administration of opiates alone is without effect on ileus.

Postoperative ileus is largely inflammatory in origin, and appears to be reduced when surgical techniques (e.g. minimally invasive approaches) are used that are associated with less inflammatory responses (as determined from interleukin-6 and C-reactive protein levels). The observation that non-steroidal anti-inflammatory drugs are effective in reducing the duration of ileus supports this hypothesis (but these are often avoided because of concern for bleeding).

Taken together, these findings suggest that epidural analgesia with local anesthetics may shorten the duration of postoperative ileus because of an anti-inflammatory action of the local anesthetic. Modulating effects of local anesthetics on the inflammatory system are well known, and have been described in vitro, in animal studies, and to a lesser extent in clinical trials. In animals, inflammatory-mediated injury in heart is ameliorated by local anesthetics, as is endotoxin- or acid-mediated lung injury. In humans, thrombosis incidence11 and hypercoagulation after surgery (both inflammatory-mediated processes) are decreased by systemic local anesthetics (yet physiologic coagulation is not affected). Important in the current context, the effectiveness of local anesthetics in the setting of inflammatory bowel disease is well established. The compounds have been shown to decrease the release of inflammatory mediators from neutrophils, which may play a role in this beneficial effect. As another example, cognitive deficits after cardiac surgery probably result from a combination of emboli and the inflammatory response that these induce in the brain. Systemic local anesthetics would be expected to interfere with both of these processes, and indeed improve cognitive outcome in this setting.16 The mechanism behind this action is most likely a modulatory effect of local anesthetics on neutrophils. Local anesthetics have been shown to inhibit neutrophil priming (a critical component of neutrophil-mediated tissue injury), but not to interfere with activation (required for wound healing and host defense). Importantly, and in contrast to classic inflammatory suppression, this inflammatory modulation by local anesthetics is therefore not associated with detrimental effects on wound healing and infection rates. We have shown that selective inhibition by local anesthetics of cellular Gq proteins explains this effect. Other effects, including those on mediator release, may also play a role. Since epidural anesthesia leads to significant blood levels of local anesthetics (1 to 5 µM), it is conceivable that the inflammatory modulatory action of systemically absorbed local anesthetic explains the beneficial effects of epidural analgesia on duration of postoperative ileus. An additional beneficial effect on return of bowel function will result from the reduced requirement for opiate analgesics.

If this is the case, then a similar beneficial effect might be obtained using systemic administration of local anesthetics. Both the inflammatory modulatory effects and the analgesic actions (thereby decreasing opiate requirements) are present when these drugs are given intravenously. This approach would have significant advantages over epidural administration. The common use of perioperative anticoagulation for the prevention of deep venous thrombosis has made appropriate timing of epidural placement and removal considerably more difficult. Epidural placement and management costs time and adds expense. Many patients may not desire the placement of an epidural catheter. In addition, the uncommon but real risks of epidural placement (certainly in the thoracic region) would be avoided by systemic administration of the local anesthetic. The major risks are epidural hematoma or abscess, both of which can be devastating.

Several clinical trials indicate that systemic local anesthetics have beneficial actions on the return of bowel function after surgery. In patients undergoing radical prostatectomy, administration of lidocaine (3 mg/min) for the duration of surgery and 1 h postoperatively resulted in a 1 day earlier return of bowel function and an associated earlier discharge from the hospital as compared with placebo. Significantly earlier return of propulsive motility in the colon was also observed in patients undergoing cholecystectomy who received intravenous lidocaine (3 mg/min intraoperatively and continued 24 h post surgery). Similarly, intraoperative instillation of bupivacaine demonstrated beneficial effects on colonic motility.

However, no study has investigated the effect on postoperative bowel function of systemically administered local anesthetic after bowel surgery. It is in this setting that restoration of bowel function is most relevant. We hypothesize that intravenous, intraoperative and postoperative administration of local anesthetic, added to patient-controlled analgesia (PCA) for post-operative pain relief, will result in more rapid return of bowel function as compared with PCA alone. This hypothesis will be tested in a randomized, blinded, controlled clinical trial in patients undergoing open colectomy for tumor.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Scheduled for colon tumor resection.
* American Society of Anesthesiologists (ASA) physical classification classes I, II, and III.

Exclusion Criteria:

* Age <18 or >75 years
* Allergy to local anesthetics
* Severe cardiovascular disease (myocardial infarction within 6 months, profoundly decreased left ventricular function (ejection fraction <40%), or high-grade arrhythmias) or liver disease (known AST or ALT or bilirubin >2.5 times the upper limit of normal)
* Systemic corticosteroid use
* Chronic use of opiates
* Unwillingness or contraindication to epidural analgesia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
time from end of surgery to first sign of bowel function (stool or flatus) | follow-up after surgery

SECONDARY OUTCOMES:
Postoperative pain and opiate consumption | post-surgery follow-up
postoperative nausea and antiemetic use | post-surgery follow-up
duration of hospital stay | post-surgery follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marcel E Durieux, MD PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Swenson BR, Gottschalk A, Wells LT, Rowlingson JC, Thompson PW, Barclay M, Sawyer RG, Friel CM, Foley E, Durieux ME. Intravenous lidocaine is as effective as epidural bupivacaine in reducing ileus duration, hospital stay, and pain after open colon resection: a randomized clinical trial. Reg Anesth Pain Med. 2010 Jul-Aug;35(4):370-6. doi: 10.1097/AAP.0b013e3181e8d5da. PMID 20588151